CLINICAL TRIAL: NCT04111341
Title: A Double Blind, Randomized, Placebo Controlled Clinical Trial to Evaluate the Safety and Efficacy of Traditional Chinese Medicine in Sjögren's Syndrome.
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of Traditional Chinese Medicine in Sjögren's Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Cheng-Chung Wei, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CS16051
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Sjögren's Syndrome
Keywords: Sjögren's syndrome; Traditional Chinese Medicine; Herbs; Clinical trial; Gan-Lu-Yin; Jia-wei-Xiao-yao-San; Ye-Jiao-Teng; Suan-Zao-Ren
MeSH Terms: conditions — Sjogren's Syndrome | interventions — gan-lu-siao-du-yin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM Gan-Lu-Yin (GLY) (Experimental): TCM Gan-Lu-Yin 6g in the morning TCM Jia-Wei-Xiao-Yao-San, Ye-Jiao-Teng, Suan-Zao-Ren 8g in the evening for 12 weeks
  Interventions: Drug: TCM (Gan-Lu-Yin)GLY
- PLACEBO (Placebo Comparator): TCM Placebo 6g in the morning TCM Placebo 8g in the evening for 12 weeks
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: TCM (Gan-Lu-Yin)GLY — TCM Gan-Lu-Yin 6g in the morning TCM Jia-Wei-Xiao-Yao-San, Ye-Jiao-Teng, Suan-Zao-Ren 8g in the evening for 12 weeks
  Other Names: Gan-Lu-Yin
  Arms: TCM Gan-Lu-Yin (GLY)
Drug: PLACEBO — TCM Placebo 6g in the morning TCM Placebo 8g in the evening for 12 weeks
  Arms: PLACEBO

SUMMARY:
To investigate the efficacy and safety of traditional Chinese medicine in patients with Sjogren's syndrome.

DETAILED DESCRIPTION:
This is 2 years' double blind, randomized, placebo-controlled clinical trial. Patients fulfilled the classification criteria of Sjogren syndrome will be recruited. Eligible subjects will be randomized on a 2:1 ratio to Traditional Chinese Medicine (TCM) granules or placebo for 12 weeks. The treatment group will receive a combination formula with traditional Chinese medicine, Gan-Lu-Yin in the morning and Jia-wei-Xiao-yao-San in the evening. Primary endpoint is the ESSPRI, European Sjogren Syndrome Patient Reported Outcome Index. Secondary endpoints include disease activity index (ESSDAI) , patient global assessment (PGA), VAS pain scale, Quality of Life by Short Form-36 (SF-36), fatigue scale and related serological markers. Thirty patients will be enrolled in the first year. After interim analysis at the end of first year, sample size will be recalculated base on the interim analysis results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old
* Written informed consent obtained
* Been diagnosed with the diagnostic criteria for Sjogren's syndrome (according to the 2002 European Classification Standard)
* The ESSPRI score of the patient of Sjogren's syndrome at least> 3

Exclusion Criteria:

* Have association disease about heart, lung, nerve or mental
* Pregnant or breastfeeding women
* Laboratory abnormality:

  1. Serum creatinine ≥2.0 mg/dl
  2. Male: Hb≤9 g/dl;Female: Hb≤8.5 g/dl
  3. Neutrophil or lymphocyte<0.5 x 109/l

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) at week 12 | week 0, week 12
  The investigators use ESSPRI to compared the difference between the week 12 and 0

SECONDARY OUTCOMES:
Change from baseline EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) at week 4 | week 0, week 4
  The investigators use ESSDAI to compared the difference between the the week 4 and 0
Physicians Global Assessment to measure quality of life (PGA) | week 0, week 4, week 8, week 12
  The investigators use PGA to compared the difference between the week 12 and 0, the week 8 and 0, the week 4 and 0
Visual Analog Scale for pain (VAS) | week 0, week 4, week 8, week 12
  The investigators use VAS to compared the difference between the week 12 and 0, the week 8 and 0, the week 4 and 0
Quality of life by SF-36 | week 0, week 4, week 8, week 12
  The investigators use SF-36 to compared the difference between the week 12 and 0, the week 8 and 0, the week 4 and 0
modified fatigue impact scale (MFI) | week 0, week 4, week 8, week 12
  The investigators use MFI to compared the difference between the week 12 and 0, the week 8 and 0, the week 4 and 0
Pittsburgh Sleep Quality Index (PSQI) | week 0, week 4, week 8, week 12
  The investigators use PSQI to compared the difference between the week 12 and 0, the week 8 and 0, the week 4 and 0
Body Constitution Questionnaire (BCQ) | week 0, week 4, week 8, week 12
  The investigators use BCQ to compared the difference between the week 12 and 0, the week 8 and 0, the week 4 and 0
Change from baseline EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) at week 8 | week 0, week 8
  The investigators use ESSDAI to compared the difference between the week 8 and 0

CONTACTS AND LOCATIONS:
Overall Officials: Wei C- C, M, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No